CLINICAL TRIAL: NCT05295511
Title: Dose-response Effects of a Recreational Team Handball-based Exercise Programme on Cardiovascular, Metabolic, Musculoskeletal and Physical Fitness Markers in Inactive Middle-aged and Older Male
Brief Title: Effects of a Recreational Team Handball-based Programme on Health and Physical Fitness of Middle-aged and Older Men
Acronym: (H4HM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Collaborators: Research Center in Sports Sciences, Health Sciences and Human Development (Other); Universidade do Porto (Other); Centre of Research, Education, Innovation and Intervention in Sport, University of Porto (Unknown); University of Southern Denmark (Other); Porto Sports Medicine Center (IPDJ, IP) (Unknown); Gaia City Hall (Unknown); Portuguese Handball Federation (Unknown); São João University Hospital Centre (Unknown); EPIUnit, Public Health Institute, University of Porto (Unknown)
Responsible Party: Principal Investigator, Susana Cristina Araújo Póvoas, Associate Professor, University Institute of Maia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEFADE 19 2019
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Healthy Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Team Handball 1 (Experimental): Team handball group participants were instructed to perform one weekly 60-min recreational team handball training sessions for 16 weeks.
  Interventions: Other: Recreational Team Handball programme
- Team Handball 2 (Experimental): Team handball group participants were instructed to perform two weekly 60-min recreational team handball training sessions for 16 weeks.
  Interventions: Other: Recreational Team Handball programme
- Team Handball 3 (Experimental): Team handball group participants were instructed to perform three weekly 60-min recreational team handball training sessions for 16 weeks.
  Interventions: Other: Recreational Team Handball programme
- Control Group (No Intervention): The control group participants were instructed to keep their regular daily physical activity for 16 weeks.

INTERVENTIONS:
Other: Recreational Team Handball programme — All training sessions consisted of a standardized 15-min warm-up (running, coordination, strength, flexibility and balance exercises), followed by 3x15-min periods of recreational team handball matches interspersed by 2-min breaks, performed in an indoor team handball court. The matches were played as small and formal game formats (4v4, 5v5, 6v6 or 7v7).
  Arms: Team Handball 1; Team Handball 2; Team Handball 3

SUMMARY:
The present study aims at analyzing the dose-response effects of a recreational team handball-based exercise programme on cardiovascular, metabolic, musculoskeletal and physical fitness markers of inactive middle-aged and older men, without previous experience with the sport. The researchers hypothesized a positive weekly training frequency effect on health and physical fitness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male participants; inactive with 50 or more years of age (i.e., not complying with the physical activity guidelines for the last 6 months).

Exclusion Criteria:

* Any medical contraindication to perform moderate-to-vigorous physical activity; incapacity to run or grip a ball.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Middle-aged and older men
Enrollment: 68 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in maximal oxygen uptake | Baseline and week 16
  Maximal oxygen uptake (mL/min/kg) was measured by pulmonary gas exchange measurements. The participants performed an incremental treadmill test until voluntary exhaustion in a laboratory, according to a standardized incremental protocol.

SECONDARY OUTCOMES:
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in systolic blood pressure | Baseline and week 16
  Systolic blood pressure (mmHg) was measured in a laboratory by an automatic upper arm blood pressure monitor (multiparameter patient monitor, Omron Z207, Kyoto, Japan) according to standardized procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in diastolic blood pressure | Baseline and week 16
  Diastolic blood pressure (mmHg) was measured in a laboratory by an automatic upper arm blood pressure monitor (multiparameter patient monitor, Omron Z207, Kyoto, Japan) according to standardized procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in resting heart rate | Baseline and week 16
  Resting heart rate (bpm) was measured in a laboratory by an automatic upper arm blood pressure monitor (multiparameter patient monitor, Omron Z207, Kyoto, Japan) according to standardized procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in whole-body mass | Baseline and week 16
  Whole-body mass was measured by a whole-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in left arm total mass | Baseline and week 16
  Left arm total mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in right arm total mass | Baseline and week 16
  Right arm total mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in left leg total mass | Baseline and week 16
  Left leg total mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in right leg total mass | Baseline and week 16
  Right leg total mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in gynoid total mass | Baseline and week 16
  Gynoid total mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in android total mass | Baseline and week 16
  Android total mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in whole-body fat mass | Baseline and week 16
  Whole-body fat mass was measured by a whole-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in left arm fat mass | Baseline and week 16
  Left arm fat mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in right arm fat mass | Baseline and week 16
  Right arm fat mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in left leg fat mass | Baseline and week 16
  Left leg fat mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in right leg fat mass | Baseline and week 16
  Right leg fat mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in gynoid fat mass | Baseline and week 16
  Gynoid fat mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in android fat mass | Baseline and week 16
  Android fat mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in whole-body lean mass | Baseline and week 16
  Whole-body lean mass was measured by a whole-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in left arm lean mass | Baseline and week 16
  Left arm lean mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in right arm lean mass | Baseline and week 16
  Right arm lean mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in left leg lean mass | Baseline and week 16
  Left leg lean mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in right leg lean mass | Baseline and week 16
  Right leg lean mass was measured by a regional-body dual- energy X-ray absorptiometry following standard procedures
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in whole-body bone mineral density | Baseline and week 16
  Whole-body bone mineral density dual- energy X-ray absorptiometry scans following standard procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in whole-body bone mineral content | Baseline and week 16
  Whole-body bone mineral content dual- energy X-ray absorptiometry scans following standard procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in lumbar spine bone mineral density | Baseline and week 16
  Lumbar spine bone mineral density dual- energy X-ray absorptiometry regional scans following standard procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in lumbar spine bone mineral content | Baseline and week 16
  Lumbar spine bone mineral content dual- energy X-ray absorptiometry regional scans following standard procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in femur bone mineral density | Baseline and week 16
  Femur bone mineral density dual- energy X-ray absorptiometry regional scans following standard procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in femur bone mineral content | Baseline and week 16
  Femur bone mineral content dual- energy X-ray absorptiometry regional scans following standard procedures.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in procollagen type-1 amino-terminal propeptide | Baseline and week 16
  Plasma concentrations of biochemical bone turnover markers were analyzed by chemiluminescence method using a fully automated immunoassay system.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in osteocalcin | Baseline and week 16
  Plasma concentrations of biochemical bone turnover markers were analyzed by chemiluminescence method using a fully automated immunoassay system.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in carboxy-terminal type-1 collagen crosslinks | Baseline and week 16
  Plasma concentrations of biochemical bone turnover markers were analyzed by chemiluminescence method using a fully automated immunoassay system.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in sclerostin | Baseline and week 16
  Plasma concentrations of biochemical bone turnover markers were analyzed by chemiluminescence method using a fully automated immunoassay system.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in isometric upper body strength | Baseline and week 16
  Isometric upper body strength was measured by a handgrip dynamometer (kg).
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in postural balance | Baseline and week 16
  Postural balance was evaluated by the number of falls in a single-legged flamingo balance test.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in upper and lower body strength, and coordination | Baseline and week 16
  Upper and lower body strength (N), and coordination (s) tests were measured according to Rikili and Jones ( 2013) standardized protocols.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in aerobic performance | Baseline and week 16
  Aerobic performance (Yo-Yo intermittent endurance level 1 test; YYIE1) (m) was evaluated on an indoor team handball court, acording to a standardized protocol.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in total cholesterol | Baseline and week 16
  Total cholesterol (mg/dl) was determined by an automated analyzer.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in high-density lipoprotein cholesterol | Baseline and week 16
  High-density lipoprotein cholesterol (mg/dl) was determined by an automated analyzer.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in low-density lipoprotein cholesterol | Baseline and week 16
  Low-density lipoprotein cholesterol (mg/dl) was determined by an automated analyzer.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in triglycerides | Baseline and week 16
  Triglycerides (mg/dl) was determined by an automated analyzer.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in glycosylated haemoglobin | Baseline and week 16
  Glycosylated haemoglobin (%) was determined by an automated analyzer.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in glucose | Baseline and week 16
  Glucose (mg/dl) was determined by an automated analyzer.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in insulin | Baseline and week 16
  Fasting blood insulin (µmol/L) was determined was determined by an automated analyzer.
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in total antioxidant status | Baseline and week 16
  Total antioxidant status (TAS) (mmol/L) was measured in plasma samples using AU5800 (Beckman-Coulter®, USA)
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in glutathione reductase | Baseline and week 16
  Glutathione reductase (GR) (U/L) was measured in plasma samples using AU5800 (Beckman-Coulter®, USA)
Within-group changes from baseline to 16 weeks, and between-group changes in week 16, in glutathione peroxidase | Baseline and week 16
  Glutathione peroxidase (GPx) (U/L) was measured in plasma samples using AU5800 (Beckman-Coulter®, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Póvoas, Principal Investigator — University of Maia
Locations (1):
- Univerisity of Maia, Maia, Porto District, Portugal

REFERENCES:
- [Derived] Carneiro I, Krustrup P, Castagna C, Pereira R, Jorgensen NR, Coelho E, Povoas S. Bone health, body composition and physical fitness dose-response effects of 16 weeks of recreational team handball for inactive middle-to-older-aged males - A randomised controlled trial. Eur J Sport Sci. 2023 Nov;23(11):2251-2263. doi: 10.1080/17461391.2023.2222685. Epub 2023 Jul 10. PMID 37376804
- [Derived] Carneiro I, Krustrup P, Castagna C, Mohr M, Magalhaes J, Pereira R, Santos R, Martins S, Guimaraes JT, Coelho E, Povoas S. Dose-response effect of a recreational team handball-based exercise programme on cardiometabolic health and physical fitness in inactive middle-aged-to-elderly males - a randomised controlled trial. Eur J Sport Sci. 2023 Nov;23(11):2178-2190. doi: 10.1080/17461391.2023.2213195. Epub 2023 Jul 19. PMID 37162301